CLINICAL TRIAL: NCT02039414
Title: Effects of Physical Activity on Maternal Lipid Metabolism, Oxidative Stress, and Neonatal Outcomes in Obese Pregnancy
Brief Title: Effects of Obesity and Physical Inactivity on Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201306109; TL1TR000449 (NIH)
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Sedentary
Keywords: Obesity; Physical Inactivity; Lipid Oxidation; Oxidative stress; pregnancy; neonatal adiposity; neonatal insulin sensitivity
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The investigators are collecting maternal blood at 7 different time points (all in one day/visit) during the 3rd trimester of thier pregnancy. The investigators are also collecting cord blood when the babies are born. All of these samples are stored at -80 with patient identification numbers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese, Inactive: Pregnant women with a BMI≥30kg/m2 and sedentary lifestyle
- Obese, Active: Pregnant women with a BMI≥30kg/m2 and exercising >150min/week

SUMMARY:
Regular maternal physical activity leads to the delivery of lighter, leaner infants. Higher birth weights and childhood obesity are both strong predictors for adult obesity, suggesting that the impact of maternal physical activity on the future health of a child is substantial. However, the mechanisms underlying the relationships between maternal physical activity and improved infant outcomes are unclear. Thus, the purpose of this project is to measure two potential contributing factors: maternal fat metabolism and maternal oxidative stress profiles. The investigators believe that maternal physical activity leads to beneficial alterations in maternal fat metabolism and oxidative stress profiles. Further, the investigators believe that both maternal fat metabolism and oxidative stress levels are related to infant outcomes such as obesity and insulin resistance. Therefore, exercise will improve maternal metabolic factors that can lead to improvements in infant outcomes. The investigators will compare these factors between obese inactive pregnant women and obese active pregnant women. This study design will allow us not only to determine the effect of physical activity on maternal and neonatal pregnancy outcomes, but also to establish whether obesity or physical inactivity should be a primary area of focus when prescribing pregnancy interventions in clinical practice.

DETAILED DESCRIPTION:
Exercise during pregnancy is associated with the delivery of leaner, lighter, and healthier infants (Clapp 1990, Clapp 2000). Subsequently, high infant adiposity and birth weight are strong predictors of childhood obesity and adult adiposity (Catalano 2006, Danielzk 2002). Therefore, maternal physical inactivity during pregnancy may have significant ramifications for the child, the effects of which may extend well into adulthood. Exercise during pregnancy also plays an important role in the health of the mother. Active pregnant women tend to gain less weight during pregnancy (Clapp 1995) and retain less weight following pregnancy (O'Toole, 2003). With excessive gestational weight gain being the strongest risk factor for maternal overweight and obesity postpartum, as well as being associated with many adverse maternal and neonatal metabolic outcomes such as adiposity and insulin resistance (Heerwagen 2010), the impact of exercise on maternal and neonatal outcomes could be substantial. The mechanisms underlying these changes are poorly understood and studies which strive to expose them are critical.

Habitual physical activity in non-gravid individuals has been shown to positively alter lipid metabolism by increasing fatty acid oxidation (Martin 1996), but the effect of physical activity on maternal lipid metabolism during pregnancy has not been studied. Due to previous research suggesting that an altered intrauterine metabolic environment may play a significant role in fetal programming (Heerwagen 2010), it is reasonable to believe improvements in maternal lipid metabolism may contribute to improved neonatal metabolic outcomes in exercising pregnant women. Preliminary data from our group found that in obese and lean pregnant women, lipid oxidation rate was significantly correlated to offspring birth weight; suggesting maternal lipid metabolism may contribute to neonatal metabolic outcomes. In inactive pregnant women, impaired lipid oxidative capacity in conjunction with known increased physiologic adipose tissue lipolysis that occurs during pregnancy and obesity would result in excess un-oxidized plasma fatty acids that are likely to be re-esterified in adipose tissue and/or delivered to the fetus. This series of events may contribute to increased maternal and neonatal adiposity.

In addition, generation of excess reactive oxygen species, known byproducts of lipid metabolism, may contribute to altered/abnormal oxidative stress profiles in obese pregnant women. Reactive oxygen species are up-regulated during physiologic pregnancy as well as non-gravid obesity, and research suggests oxidative stress may be related to poorer neonatal outcomes (Heerwagen 2010) . In non-gravid individuals, long-term physical activity has been shown to improve oxidative stress profiles (Fisher-Wellman 2009). Therefore, women who exercise during pregnancy may also have higher antioxidant capacity and lower markers of oxidative stress; both of which may contribute to favorable neonatal outcomes. However, this has not yet been studied.

Obesity is also believed to adversely influence lipid metabolism, oxidative stress, and neonatal outcomes in pregnancy. Therefore, we plan to compare these parameters in obese active and obese inactive pregnant women. This study design will allow us to compare groups in order to determine if unfavorable maternal lipid metabolism and oxidative stress profiles, and neonatal metabolic outcomes (adiposity and insulin resistance) are more attributable to physical inactivity or obesity. Previous research with non-gravid adults suggests that the presence of comorbidity is more correlated with physical activity levels than with body weight (Blair 1989, 1999, Sui 2007). This finding is contrary to much of the previous literature on pregnancy which suggests "obesity may be the most common health risk for the developing fetus" (Heerwagen 2010). Knowledge about maternal lipid metabolism and oxidative stress profiles and their relationships in neonatal outcomes in active and inactive pregnant women can guide lifestyle and medical interventions designed to target factors that may be contributing to poor outcomes in obese pregnancy. Currently, we have collected data on lean, inactive pregnant women that can be used for comparison at the end of all data collection.

This is the first study to examine the relationship between physical activity, lipid metabolism and oxidative stress in obese pregnancy. We anticipate that results from the proposed study will demonstrate the importance of a physically active lifestyle during pregnancy (irrespective of body weight) in order to maximize the short and long-term health of the neonate. In addition, we hope that these results will encourage obese and overweight women of childbearing age to remain or become physically active by demonstrating that physical inactivity has a greater effect on poor neonatal outcomes than obesity. These findings are unique as much of the current literature focuses on the negative impact of maternal obesity on neonatal outcomes. Blair et al. has consistently demonstrated in non-gravid populations that physical inactivity is a stronger predictor of all-cause mortality than obesity (Blair 1989, 1999). Similarly, we believe physical activity in pregnancy is more important than simply maintaining a healthy body weight in improving neonatal outcomes. This idea is novel and innovative as it is previously unexplored in pregnancy and pregnancy outcomes.

In addition to determining the effect of regular physical activity on neonatal outcomes, measuring maternal lipid metabolism and oxidative stress profiles will provide valuable knowledge about mechanisms responsible for improved outcomes in physically active pregnant women. Also, measuring maternal lipid metabolism and oxidative stress profiles during exercise is novel and clinically insightful. This paradigm holds the potential to reveal alterations in maternal metabolism and/or oxidative stress profiles that may not be detected when measuring these factors at rest. Additionally, measuring metabolism and oxidative stress during exercise is clinically useful by providing information about maternal metabolism during activities that will mimic daily lifestyle tasks such as childcare, household chores, etc. (~3-5 METS). Thus, this study design will provide us with valuable insight and enhanced understanding of maternal lipid metabolism and oxidative stress profiles during everyday lifestyle activities.

METHODS

Subjects:

All women who seek pre-natal care at the Women's Health Clinic at Barnes Jewish Hospital/Washington University will be screened for inclusion BMI by history at the clinic. Subjects will be recruited late in their 2nd trimester at the women's health clinic after asking about their exercise habits. All patients who meet criterion with on-going pregnancies will be approached for enrollment in the study. This study will compare 2 groups of pregnant women between 30 and 35 weeks gestation. The first group will inactive obese women and the other will be active obese women. We will recruit ~15 subjects per group (N=30). Groups will be race-matched.

Sample Size Calculation Data from Pomeroy et al.in 2012 stated that when using an accelerometer to measure physical activity and air displacement plethysmography to measure neonatal body composition (the same measurements we are proposing to use), the Spearman correlation coefficient showing the association between maternal physical activity level and neonatal fat free mass is r=0.5226. Using this R-value and an alpha of 0.05, 30 total participants (15 per group) are needed to adequately power our study at .85 (beta=.15).

Study Procedures:

All study procedures will be performed at the Washington University School of Medicine (WUSM) Institute for Clinical and Translational Sciences Clinical Research Unit (CRU).

CRU Visit #1 of 2: Body composition and Fitness Assessment (32-37 weeks gestation):

Maternal Body Composition:

A skin fold measurement will be performed to determine maternal body composition (% body fat). This will be done by pressing folds of the skin at 7 sites with a caliper and recording its thickness as previously described (Jackson and Pollock 1980).

Maternal Physical Fitness Levels:

Maternal fitness levels will be assessed using a submaximal cycle test on a recumbent bicycle. Subjects will sit comfortably on the bicycle while the pedals are properly adjusted so there is a slight bend in the knee when legs are extended. They will then complete the YMCA submaximal multistage cycle ergometer test according ACSM's guidelines for exercise testing and prescription (Thompson 2010). Sady and colleagues concluded that the VO2-Heart Rate extrapolation method is the most precise way to predict VO2max in pregnancy (1985)., and the YMCA test utilizes this method. A 3-lead ECG will be applied to monitor heart rate during the exercise test.

Maternal Physical Activity Levels:

Daily maternal physical activity will be assessed in the week following these tests using the ActiGraph GT3X+ accelerometer (ActiGraph LLC, Pensacola, FL) in order to objectively measure daily physical activity levels. ActiGraph data will be collected for seven consecutive days on the non-dominant wrist at 30 Hertz. Time spent in sedentary and active (light, lifestyle, moderate, vigorous, and very vigorous) activities will be calculated using algorithms from Freedson and colleagues using ActiGraph software (Freedson 1998). We will also measurement maternal physical activity levels subjectively using the Pregnancy Physical Activity Questionnaire (PPAQ). The PPAQ is a valid and reliable instrument to measure physical activity levels during pregnancy (Chasan-Taber 2011). Not only will the PPAQ provide us with additional details about their activity levels, but it will allow us to account for activities that the actigraph may be unable to detect (i.e. riding a stationary bicycle).

Dietary Intake and Composition:

In order to account for differences in diet, subjects will complete the National Institutes of Health's Dietary History Questionnaire II. This dietary assessment has been rigorously validated (Subar 2001) and is widely used among many different populations. Previous literature also demonstrates that dietary history questionnaires are valid and reproducible among pregnant populations (Vioque 2013).

CRU Visit #2 of 2: Lipid metabolism during exercise study (32-37 weeks gestation):

After obtaining height, weight, and vitals, a catheter (IV) will be placed in a hand vein and heated in a warming box prior to each blood draw. Participants will rest for approximately 30 minutes prior to measuring lipid oxidation rate using indirect calorimetry (True One 2400, Parvo Medics, Sandy, UT). Participants will lay supine while a hood device is placed over their head for 15 minutes to measure oxygen consumption and carbon dioxide production in order to determine lipid oxidation rate34. After the initial indirect calorimetry measurement is taken, basal blood collection will be obtained. Basal insulin and glucose levels will be used to calculate maternal insulin resistance via a homeostatic model assessment-insulin resistance (HOMA-IR). After this blood draw, participants will exercise at approximately 50% of their predicted VO2max (based on the YMCA submaximal cycle test) for 30 minutes on the recumbent cycle ergometer (Lode Corvial, InMed, New South Wales, Australia). Blood will be collected at various time points during exercise. Indirect calorimetry (using a mouthpiece, nose clip, and exercise version of the software) will also be performed for 2 minutes at a time to measure lipid oxidation and total body oxygen consumption during low-level exercise. After exercise termination, participants will return to a supine position. Recovery blood draws will be taken and indirect calorimetry will be performed.

Blood drawn at different time points will be used to measure glucose, insulin, free fatty acids, reactive oxygen species (F2- isoprostanes by mass spectrometry (also referred to as 8-iso-PGF2α) (Milne 2007)), and total antioxidant capacity (Total Antioxidant Capacity Assay (TAC), Cell Biolabs, Inc., San Diego, CA). All of these measurements will help us to better understand insulin resistance, oxidative stress, and mechanisms that could be contributing to either condition.

Parturition:

At parturition, maternal weight will be measured and gestational weight gain will be determined. Neonatal weight, length, and head circumference will also be obtained. Infant HOMA-IR and fatty acid delivery to the fetus will be determined by measuring umbilical cord plasma glucose, insulin, and fatty acid concentrations at parturition. Within 48 hours of delivery, neonatal body composition (fat and lean mass) will be measured by skin fold thickness measurement and by air displacement plethysmography (Pea Pod, Life Measurement, Inc., Concord, CA) in the CRU at WUSM.

Statistical Analysis: Repeated measures ANOVA (group x time) will be used to compare lipid oxidation rates and oxidative stress profiles between the 2 groups during pregnancy before, during, and after exercise. Pearson product moment correlation coefficients for normally distributed variables and Spearmen's rank order coefficients for non-normally distributed variables will be used to examine the relationships between maternal lipid oxidation rate, plasma oxidative stress markers, and neonatal metabolic outcomes. We may also use a regression analysis to examine the relationship between maternal physical activity levels in obese women and neonatal body composition and/or insulin resistance (similar to what has been done in normal weight pregnant women by Pomeroy et al. 2012).

ELIGIBILITY:
Inclusion Criteria:

* . Age 18-44 2. Confirmed singleton viable pregnancy with no fetal abnormalities at routine 18-22 ultrasonography 3. Obese: Pre-pregnancy BMI between 30 and 45 kg/m2 4. Receipt of prenatal care and plans to deliver at Barnes-Jewish Hospital 5. Inactive: < 30min of low intensity activity (>1.5 METS) all or most days of the week Physically Active: >150 minutes/week of moderate to high intensity activity 6. Completion of a normal routine, standard of care 1 hour 50 gram gestational diabetes screen

Exclusion Criteria:

1. Multiple gestation pregnancy
2. Inability to provide voluntary informed consent
3. Current use of illegal drugs (cocaine, methamphetamine, opiates, etc…)
4. Current smoker who does not consent to cessation
5. Current usage of daily medications by class: corticosteroids, anti-psychotics (known to alter insulin resistance and metabolic profiles)
6. History of gestational diabetes, pre-pregnancy diabetes or prior macrosomic (>4500g) infant (each elevate the risk for gestational diabetes in the current pregnancy, or undiagnosed gestational diabetes)
7. History of heart disease.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women who seek pre-natal care at the Women's Health Clinic at Barnes Jewish Hospital/Washington University will be screened for inclusion BMI by history at the clinic. Subjects will be recruited late in their 2nd trimester at the women's health clinic after asking about their exercise habits. All patients who meet criterion with on-going pregnancies will be approached for enrollment in the study. This study will compare 2 groups of pregnant women between 32 and 37 weeks gestation. The first group will inactive obese women and the other will be active obese women. We will recruit 15 subjects per group (N=30). Groups will be race-matched.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Cade, PT, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Clapp JF 3rd, Dickstein S. Endurance exercise and pregnancy outcome. Med Sci Sports Exerc. 1984 Dec;16(6):556-62. PMID 6513772
- [Background] Clapp JF 3rd. The course of labor after endurance exercise during pregnancy. Am J Obstet Gynecol. 1990 Dec;163(6 Pt 1):1799-805. doi: 10.1016/0002-9378(90)90753-t. PMID 2256485
- [Background] Clapp JF 3rd, Capeless EL. Neonatal morphometrics after endurance exercise during pregnancy. Am J Obstet Gynecol. 1990 Dec;163(6 Pt 1):1805-11. doi: 10.1016/0002-9378(90)90754-u. PMID 2256486
- [Background] Clapp JF 3rd, Little KD. Effect of recreational exercise on pregnancy weight gain and subcutaneous fat deposition. Med Sci Sports Exerc. 1995 Feb;27(2):170-7. PMID 7723638
- [Background] Clapp JF 3rd. Exercise during pregnancy. A clinical update. Clin Sports Med. 2000 Apr;19(2):273-86. doi: 10.1016/s0278-5919(05)70203-9. PMID 10740759
- [Background] Clapp JF 3rd. Long-term outcome after exercising throughout pregnancy: fitness and cardiovascular risk. Am J Obstet Gynecol. 2008 Nov;199(5):489.e1-6. doi: 10.1016/j.ajog.2008.05.006. Epub 2008 Jul 29. PMID 18667190
- [Background] Magann EF, Evans SF, Weitz B, Newnham J. Antepartum, intrapartum, and neonatal significance of exercise on healthy low-risk pregnant working women. Obstet Gynecol. 2002 Mar;99(3):466-72. doi: 10.1016/s0029-7844(01)01754-9. PMID 11864675
- [Background] Danielzik S, Langnase K, Mast M, Spethmann C, Muller MJ. Impact of parental BMI on the manifestation of overweight 5-7 year old children. Eur J Nutr. 2002 Jun;41(3):132-8. doi: 10.1007/s00394-002-0367-1. PMID 12111051
- [Background] Demerath EW, Reed D, Rogers N, Sun SS, Lee M, Choh AC, Couch W, Czerwinski SA, Chumlea WC, Siervogel RM, Towne B. Visceral adiposity and its anatomical distribution as predictors of the metabolic syndrome and cardiometabolic risk factor levels. Am J Clin Nutr. 2008 Nov;88(5):1263-71. doi: 10.3945/ajcn.2008.26546. PMID 18996861
- [Background] Heerwagen MJ, Miller MR, Barbour LA, Friedman JE. Maternal obesity and fetal metabolic programming: a fertile epigenetic soil. Am J Physiol Regul Integr Comp Physiol. 2010 Sep;299(3):R711-22. doi: 10.1152/ajpregu.00310.2010. Epub 2010 Jul 14. PMID 20631295
- [Background] Keppel KG, Taffel SM. Pregnancy-related weight gain and retention: implications of the 1990 Institute of Medicine guidelines. Am J Public Health. 1993 Aug;83(8):1100-3. doi: 10.2105/ajph.83.8.1100. PMID 8342716
- [Background] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411
- [Background] Wolff S, Legarth J, Vangsgaard K, Toubro S, Astrup A. A randomized trial of the effects of dietary counseling on gestational weight gain and glucose metabolism in obese pregnant women. Int J Obes (Lond). 2008 Mar;32(3):495-501. doi: 10.1038/sj.ijo.0803710. Epub 2008 Jan 29. PMID 18227847
- [Background] Martin WH 3rd. Effects of acute and chronic exercise on fat metabolism. Exerc Sport Sci Rev. 1996;24:203-31. PMID 8744251
- [Background] Jarvie E, Hauguel-de-Mouzon S, Nelson SM, Sattar N, Catalano PM, Freeman DJ. Lipotoxicity in obese pregnancy and its potential role in adverse pregnancy outcome and obesity in the offspring. Clin Sci (Lond). 2010 Apr 28;119(3):123-9. doi: 10.1042/CS20090640. PMID 20443782
- [Background] Rkhzay-Jaf J, O'Dowd JF, Stocker CJ. Maternal Obesity and the Fetal Origins of the Metabolic Syndrome. Curr Cardiovasc Risk Rep. 2012 Oct;6(5):487-495. doi: 10.1007/s12170-012-0257-x. Epub 2012 Aug 14. PMID 23002417
- [Background] Herrera E. Lipid metabolism in pregnancy and its consequences in the fetus and newborn. Endocrine. 2002 Oct;19(1):43-55. doi: 10.1385/ENDO:19:1:43. PMID 12583601
- [Background] Catalano PM, Roman-Drago NM, Amini SB, Sims EA. Longitudinal changes in body composition and energy balance in lean women with normal and abnormal glucose tolerance during pregnancy. Am J Obstet Gynecol. 1998 Jul;179(1):156-65. doi: 10.1016/s0002-9378(98)70267-4. PMID 9704782
- [Background] Catalano PM, Ehrenberg HM. The short- and long-term implications of maternal obesity on the mother and her offspring. BJOG. 2006 Oct;113(10):1126-33. doi: 10.1111/j.1471-0528.2006.00989.x. Epub 2006 Jul 7. PMID 16827826
- [Background] Catalano, P. M. (2010).
- [Background] Sen, S. and R. A. Simmons
- [Background] Sui X, LaMonte MJ, Laditka JN, Hardin JW, Chase N, Hooker SP, Blair SN. Cardiorespiratory fitness and adiposity as mortality predictors in older adults. JAMA. 2007 Dec 5;298(21):2507-16. doi: 10.1001/jama.298.21.2507. PMID 18056904
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Blair SN, Brodney S. Effects of physical inactivity and obesity on morbidity and mortality: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S646-62. doi: 10.1097/00005768-199911001-00025. PMID 10593541
- [Background] Pomeroy, J., et al. (2013).
- [Background] Thompson, W.R. (2010) ACSM's Guidelines for Exercise Testing and Perscription. 8th edition. Philadelphia, PN: Lippencott Williams & Wilkins
- [Background] Jackson AS, Pollock ML, Ward A. Generalized equations for predicting body density of women. Med Sci Sports Exerc. 1980;12(3):175-81. PMID 7402053
- [Background] Sady SP, Carpenter MW, Sady MA, Haydon B, Hoegsberg B, Cullinane EM, Thompson PD, Coustan DR. Prediction of VO2max during cycle exercise in pregnant women. J Appl Physiol (1985). 1988 Aug;65(2):657-61. doi: 10.1152/jappl.1988.65.2.657. PMID 3170418
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Chasan-Taber L, Schmidt MD, Roberts DE, Hosmer D, Markenson G, Freedson PS. Development and validation of a Pregnancy Physical Activity Questionnaire. Med Sci Sports Exerc. 2004 Oct;36(10):1750-60. doi: 10.1249/01.mss.0000142303.49306.0d. PMID 15595297
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Vioque, J., et al. (2013).
- [Background] Frayn KN. Calculation of substrate oxidation rates in vivo from gaseous exchange. J Appl Physiol Respir Environ Exerc Physiol. 1983 Aug;55(2):628-34. doi: 10.1152/jappl.1983.55.2.628. PMID 6618956
- [Background] Milne GL, Yin H, Brooks JD, Sanchez S, Jackson Roberts L 2nd, Morrow JD. Quantification of F2-isoprostanes in biological fluids and tissues as a measure of oxidant stress. Methods Enzymol. 2007;433:113-26. doi: 10.1016/S0076-6879(07)33006-1. PMID 17954231
- [Background] O'Toole ML, Sawicki MA, Artal R. Structured diet and physical activity prevent postpartum weight retention. J Womens Health (Larchmt). 2003 Dec;12(10):991-8. doi: 10.1089/154099903322643910. PMID 14709187
- [Background] Fisher-Wellman K, Bell HK, Bloomer RJ. Oxidative stress and antioxidant defense mechanisms linked to exercise during cardiopulmonary and metabolic disorders. Oxid Med Cell Longev. 2009 Jan-Mar;2(1):43-51. doi: 10.4161/oxim.2.1.7732. PMID 20046644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese, Inactive | Obese, Active
Started | 22 | 18
Completed | 16 | 16
Not Completed | 6 | 2
Not completed — Delivered | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese, Inactive | Obese, Active | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.0 (4.8) | 28.9 (4.8) | 26.95 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Nulliparous [Number; unit: participants] — Nulliparous: A woman who has never borne offspring (i.e. has not had a child)
  participants | 12 | 9 | 21
Low Income [Number; unit: participants] — Women were considered low-income for this study if they were recruited from a specialized clinic that required it's patients to either be on Medicaid or have no insurance. Thus, because they qualified for Medicaid or had no insurance, they were considered low-income.
  participants | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Adiposity
Description: Within 48 hours of delivery, neonatal body composition (% fat mass) will be measured by skin fold thickness measurement and by air displacement plethysmography (Pea Pod, Life Measurement, Inc., Concord, CA) in the CRU at WUSM.
Time Frame: 24-48 hr after delivery
Population: Several babies were not able to be measured for this part of the study- the primary reason being a weekend delivery that was discharged before measurements could be obtained by the study team. Our clinical research unit was not open on weekends to the the Peapod scans. This explains why there were only 15 babies per group for this outcome.
Measure: Mean (Standard Deviation); unit: % fat
Arm/Group | Obese, Inactive | Obese, Active
Number analyzed (Participants) | 15 | 15
% fat | 11.2 (3.6) | 12.4 (2.9)

2. Primary Outcome: Neonatal Insulin Resistance
Description: Infant HOMA-IR will be determined by measuring umbilical cord plasma glucose and insulin concentrations at parturition vis cord blood collection. Cord blood will be collected within 30 min of delivery, centrifuged for 10 min at 3000rpm to remove plasma, and stored at -80.
Time Frame: Immediately after delivery
Population: We could not obtain cord blood on all infants (thus, specimens were obtained fro 14 obese active and 12 obese inactive women). Due to medical emergencies or lack-of cord blood available, there were several instances where these specimens could not be obtained by the study team.
Measure: Mean (Standard Deviation); unit: HOMA_IR, unitless measure
Arm/Group | Obese, Inactive | Obese, Active
Number analyzed (Participants) | 14 | 12
HOMA_IR, unitless measure | 1.6 (1.2) | 1.9 (1.6)

3. Secondary Outcome: Maternal Inflammation
Description: High-Sensitivity C-reactive protein was measured.
Time Frame: This was taken while fasted and under resting conditions at the beginning of visit 2 (between 32 and 37 weeks gestation). This value was only measured at baseline (i.e. one timepoint).
Population: Of the 40 women consented, only 32 (16 in each group, completed the study visits). Thus, these 32 have CRP data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Obese, Inactive | Obese, Active
Number analyzed (Participants) | 16 | 16
mg/L | 9.1 (4.0) | 6.3 (2.5)

4. Secondary Outcome: Maternal Lipid Oxidation
Description: The investigators will measure maternal lipid oxidation rate using indirect calorimetry (True One 2400, Parvo Medics, Sandy, UT) before, during, and after acute exercise. This will involve placing a hoodlike device over the subject's head as they lay supine (rest).During exercise, this involved using a mouthpiece and noseclips. Using both techniques, The investigators will be able to calculate lipid oxidation rates from the volumes of CO2 produced and volumes of O2 used.The reported measure is lipid oxidation rate during exercise. The equation used to calculate lipid oxidation is: lipid oxidation (g/min) = 1.695 VO2- 1.701 VCO2 .
Time Frame: Visit 2 (32-37 weeks gestation)- reported lipid oxidation is the average of lipid oxidation over the course of the 30min exercise bout (i.e. data collected at minutes 8-10, minutes 18-20, and minutes 28-30 of exercise, all averaged together).
Population: Of the 40 women consented, only 32 (16 per group) completed all study visits and have lipid oxidation data.
Measure: Mean (Standard Deviation); unit: g/min
Arm/Group | Obese, Inactive | Obese, Active
Number analyzed (Participants) | 16 | 16
g/min | 0.2150 (0.0864) | 0.1950 (0.0790)

ADVERSE EVENTS:
Arm/Group | Obese, Inactive | Obese, Active
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No